CLINICAL TRIAL: NCT03247244
Title: A Double-blind, Randomized, Placebo-controlled Crossover Pilot Trial of Medical Cannabis in Adults With Tourette Syndrome
Brief Title: Safety and Efficacy of Cannabis in Tourette Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment/enrollment took too long
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-7726
Record Dates: First submitted 2017-07-25; First posted 2017-08-11 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Tourette Syndrome
Keywords: Cannabis; Tics; Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome; Marijuana Abuse; Tics | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: There are four treatment schemes. All subjects will be randomized in a 1:1:1:1 ratio to one of the four treatment schemes. Participants will receive a single dose of each of the 3 cannabis products + placebo, with the order determine by their assigned treatment arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigators and analysts will be masked as to the treatment arm and product of each participant and visit. Only the pharmacists will be aware of the strain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 (Other): Three cannabis drug product formulations with different THC and CBD contents and placebo will be used in the following order: A (THC 10%, CBD <0.5%), B (THC 8.6%, CBD 8.6%), C (THC 0.6%, CBD 14%) and placebo D (THC <0.3%, CBD <0.3%).
  Interventions: Drug: Cannabis
- 2 (Other): Three cannabis drug product formulations with different THC and CBD contents and placebo will be used in the following order: B (THC 8.6%, CBD 8.6%), placebo D (THC <0.3%, CBD <0.3%), A (THC 10%, CBD <0.5%), C (THC 0.6%, CBD 14%).
  Interventions: Drug: Cannabis
- 3 (Other): Three cannabis drug product formulations with different THC and CBD contents and placebo will be used in the following order: C (THC 0.6%, CBD 14%), A (THC 10%, CBD <0.5%), placebo D (THC <0.3%, CBD <0.3%), B (THC 8.6%, CBD 8.6%).
  Interventions: Drug: Cannabis
- 4 (Other): Three cannabis drug product formulations with different THC and CBD contents and placebo will be used in the following order: placebo D (THC <0.3%, CBD <0.3%), C (THC 0.6%, CBD 14%), B (THC 8.6%, CBD 8.6%), A (THC 10%, CBD <0.5%).
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — THC 10%, CBD <0.5%
  Other Names: Marijuana
Drug: Cannabis — THC 8.6%, CBD 8.6%
  Other Names: Marijuana
Drug: Cannabis — THC 0.6%, CBD 14%
  Other Names: Marijuana

SUMMARY:
For many individuals with Tourette syndrome (TS), available medications do not help with their symptoms, or cause significant side effects. Two small controlled trials have investigated the effect of oral delta-9-tetrahydrocannabinol (THC), a principal psychoactive ingredient of cannabis, in TS patients. While these trials have shown promising results, the effect sizes were not as large and consistent as those reported by patients with regards to inhaled cannabis (smoked or vaporized). Indeed, based on anecdotal evidence, patients have much greater improvement in their symptoms using inhaled cannabis than using cannabinoid pharmaceuticals. However, there have been no controlled trials of inhaled medical cannabis for TS to date. Furthermore, various medical cannabis products are authorized in Canada with different contents of THC and cannabidiol (CBD), another primary cannabinoid. No data exists regarding the dosing, efficacy and safety of these products in the treatment of TS. To gather such data, a double-blind, randomized, crossover pilot trial will be conducted to compare the efficacy and safety of three vaporized medical cannabis products with different THC and CBD contents, as well as placebo, in adults with TS. As well, the PK/PD profile of THC and CBD of the products will be assessed and correlated with tic symptoms

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult, 18-65 years of age (inclusive) at the time of signing the informed consent.
* The subject meets current DSM-5 diagnostic criteria for TS[6], diagnosed by a neuropsychiatrist with expertise in TS and related conditions.
* YGTSS-TTS ≥16, frequency subscore = 5 and intensity subscore ≥ 2. In addition, tic free intervals do not last more than two minutes based on both self-reporting and observation by clinician at both screening and Week 0 (randomization). This requirement is for the purpose of minimizing the potential for floor effects given the relatively short window for assessing effect on symptoms in this single-dose trial.
* The subject is able and willing to refrain from using any non-study cannabis during the screening and treatment phases of the study.
* Females of childbearing potential (defined by menarche and not having undergone surgical sterilization/hysterectomy) must have a negative pregnancy test, must be practicing acceptable double-barrier methods of contraception (or can confirm abstinence at each scheduled visit), and must not be breast feeding.
* Written informed consent must be obtained from the subject prior to the initiation of any protocol-required procedures.
* The subject is able to comprehend and satisfactorily comply with the protocol requirements.

Exclusion Criteria:

* • The subject and/or his/her family have a history of psychosis, schizophrenia or bipolar disorder.

  * Sexually active females of childbearing potential who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during the trial; Females who are breast-feeding and/or who have a positive serum pregnancy test result prior at the time of screening.
  * The subject represents a significant risk of committing suicide (current suicide plan or attempt in past 2 years) or committing homicide.
  * The subject has a history of serious head injury, seizure disorder, or developmental delay (intelligence quotient≤85).
  * The subject has either of: cardiovascular disease; respiratory disease such as chronic obstructive pulmonary disease (COPD) or lung cancer (asthma is not an exclusionary criterion); hepatitis.
  * The subject has a current or past history of substance abuse within the last 5 years, with the exception of cannabis.
  * The subject is using cannabis regularly for the treatment of TS.
  * The subject has any abnormal laboratory tests and vital sign results which in the investigator's judgment is medically significant and would impact the safety of the subject or the interpretation of the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Modified Rush Video-Based Tic Rating Scale | 10 minutes
  Can be used to assess changes in frequency and severity of tics

SECONDARY OUTCOMES:
The Marijuana Effect Expectancy Questionnaire (MEEQ) | 6 hours
  To assess tolerability of cannabis products

OTHER OUTCOMES:
Area under the plasma concentration versus time curve of CBD and 11-OH-THC | 6 hours
  Determine a temporal relationship between changes in THC/CBD plasma concentrations and tic severity
Premonitory Urge for Tics Scale (PUTS) | 1 hour
  Assesses the intensity of premonitory urges
Clinical Global Impression- Improvement Scale (CGI-I) | 1 hour
  Assesses how improved symptoms are after an intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sandor, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital - Tourette Syndrome Neurodevelopmental Clinic, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Abi-Jaoude E, Bhikram T, Parveen F, Levenbach J, Lafreniere-Roula M, Sandor P. A Double-Blind, Randomized, Controlled Crossover Trial of Cannabis in Adults with Tourette Syndrome. Cannabis Cannabinoid Res. 2023 Oct;8(5):835-845. doi: 10.1089/can.2022.0091. Epub 2022 Aug 30. PMID 36040329